CLINICAL TRIAL: NCT06866067
Title: The Effect of Clip Material on the Retention of Implant Supported Mandibular Overdenture: Clinical Comparative Study
Brief Title: The Effect of Clip Material on the Retention of Implant Supported Mandibular Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Sara Medhat Mohamed Ali, Lecturer of Removable Prosthodontics, MTI University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 970/6525
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Denture Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEK clip (Other): Clip for overdenture retention made from poly-ether-ether-ketone (PEEK)
  Interventions: Device: PEEK clip
- Nylon clip (Other): Clip for overdenture retention made from nylon (C6H11NO)n
  Interventions: Device: Nylon clip

INTERVENTIONS:
Device: PEEK clip — The overdentures were attached with PEEK clip . The retention of overdenture was assessed
  Arms: PEEK clip
Device: Nylon clip — The overdentures were attached with Nylon clip . The retention of overdenture was assessed
  Arms: Nylon clip

SUMMARY:
This study is aiming to evaluate the retention of implant supported mandibular overdenture using two different clip materials namely polyoxymethylene (POM) and poly-ether-ether-ketone (PEEK) on PEEK bar at three-time intervals; immediately after placement, after 3 months and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Male.
  * Completely edentulous.
  * Age: 50-60 years.
  * Free from any systemic diseases that affect bone metabolism.
  * Good intraoral condition.
  * Anterior mandibular bone height > 13mm and width > 5mm.
  * The inter-arch space from 15mm to 17mm.

Exclusion criteria:

* Smoking and drug abusing.
* Severe maxillomandibular skeletal discrepancy.
* Bone metabolic disorders.
* History of head and neck radiotherapy.
* Intravenous bisphosphonate therapy.
* Presence of para-functional habits.
* Temporomandibular joint disorders.
* Severe bony undercuts.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — bone density
Enrollment: 12 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Overdenture retention assessed using Universal Testing Machine (Newton) | From enrollment and after 3 months and finally at the end of treatment at 6 months
  Denture resistance corresponding to vertical displacement force was obtained using a universal testing machine (INSTRON, United States) to measure retention. Each patient had his chin securely fixed on a support while seated upright. The attachment portion of the universal machine was adjusted in accordance with the device's bar being securely attached to the denture. The device gradually increased the vertical load by 10 mm per minute until the denture completely fell out of place. A tuck sound can be heard to indicate the load at the dislodgment point. Additionally, the force plot in the recorded computer software data exhibits an abrupt drop (Nexyge; Lloyd Instruments; MT-4.6). Each test was repeated five times to obtain five records, and the mean of these records was calculated. Testing was carried out on the mandibular overdenture after insertion, as well as at 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- MTI University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No